CLINICAL TRIAL: NCT05083598
Title: Wearable Health Technology for Perioperative Risk Assessment
Acronym: WELCOME
Status: Completed | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Collaborators: Politecnico di Milano (Other)
Responsible Party: Sponsor
Other Study IDs: 2881
Record Dates: First submitted 2021-10-07; First posted 2021-10-19 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Surgery--Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients undergoing major surgery: Patients aged 70 or older undergoing major non cardiac surgery, with expected surgical duration > 2 hours.
  Interventions: Other: 6 Minute walking test; Other: Frailty questionaires

INTERVENTIONS:
Other: 6 Minute walking test — The patient is asked to repetitively walk along a 15 m track, at their best speed, in six minutes. Before and after the exercise, blood arterial pressure and dyspnea level (via Borg scale) are assessed. Cardiac frequency and peripheral Oxygen saturation are assessed before the test, and every minute and in the two minutes following the exercise.
Other: Frailty questionaires — Clinical Frailty Score, Metabolic Equivalent of Task, DUKE Activity Status Index

SUMMARY:
Accurate and timely preoperative identification of high-risk patients provides opportunities to better inform and manage them. Current predictors for perioperative complications are either resource consuming or have low accuracy. The primary objective of the study is to assess if Wearable Devices may be an alternative to assess cardiopulmonary function, with low risks and lower costs.

ELIGIBILITY:
Inclusion Criteria:

* Age 70 or more
* Undergoing major non cardiac surgery
* Expected surgical duration > 2 hours.

Exclusion Criteria:

* Patients unable to express consent
* Patients undergoing urgent/emergent surgery
* Patients in which surgery is planned within less than two weeks
* Patients with limited physical activity due to limited mobility related with neurological or orthopedic disease
* Acute cardiovascular event
* Surgery conducted in locoregional anesthesia only

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients aged 70 or older undergoing major non cardiac surgery, with expected surgical duration > 2 hours.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Assess whether wearable devices (WD) can identify patients at risk for postoperative complications. | 12 months

SECONDARY OUTCOMES:
To compare performance of WD data with 6MWT, MET scale, CFS and ASA score in identifying reduced functional capacity | 24 months
A sub analysis of WD data during 6MWT will be conducted | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Humanitas Research Hospital, Rozzano, Milan, Italy

IPD SHARING:
Plan to Share IPD: No